CLINICAL TRIAL: NCT00708058
Title: Can Pacemakers, Defibrillators, and Internal Heart Failure Devices Be Used to Evaluate and Guide Management in the Emergency Department?
Brief Title: Use of Defibrillator Information in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2007H0089
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Congestive Heart Failure; Medical Device
Keywords: Implanted cardiac defibrillators; Congestive Heart Failure; Emergency Department
MeSH Terms: conditions — Heart Failure; Emergencies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study to determine the feasibility of obtaining information stored in existing Medtronic internal defibrillators in patients who present to the Emergency Department(ED) for any reason. In addition, the study will determine if this information is useful to the ED physician in managing the patient's care, specifically as it relates to heart failure.

DETAILED DESCRIPTION:
This is a prospective observational pilot study to determine if stored data regarding heart function, patient activity level, and other parameters can be used by the ED physician in order to evaluate a patient's cardiac status as it pertains to heart failure. Patients presenting to the ED and who consent have their devices interrogated by research personnel. The data is printed and provided to the treating physician who completes a brief survey about whether the data was useful in managing the patient.All subjects are contacted 30 days after ED or hospital discharge to determine if they have had any ED visits or hospital admissions during that period, and if yes, whether the visits were heart failure related. After all study procedures are performed, a team of 2 cardiologists will review the patient medical record from the study visit, as well as the data obtained from the patient's device in the ED. Each cardiologist, who will be blinded to the other's conclusion, will determine if the patient was having a heart failure exacerbation at the study visit.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* Medtronic IACD present on arrival to Emergency Dept.

Exclusion Criteria:

* minors
* prisoners
* non-Medtronic AICD
* unable to provide consent
* no telephone for 30 day follow up call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 or older who present to The Ohio State University Medical Center Emergency Department for any reason, and who have an implanted Medtronic cardiac defibrillator present
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine if Medtronic implantable device diagnostics can be used in conjunction with clinical exam to diagnose and guide Emergency Department care | During Emergency Dept. visit
To determine if there are better methods of making the device diagnostic information accessible to ED physicians/staff | During Emergency Department visit

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Hiestand, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States